CLINICAL TRIAL: NCT00313274
Title: A Double-Blind, Randomized, Parallel, Placebo-Controlled Phase III Study to Evaluate the Safety and Antiviral Activity of Clevudine (L-FMAU) 30 mg QD in Patients With HBeAg Negative Chronic Hepatitis B
Brief Title: Safety and Antiviral Activity Study of Clevudine 30 mg QD in Patients With HBeAg(-) Chronic HBV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L-FMAU-302
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2006-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine

INTERVENTIONS:
Drug: Clevudine

SUMMARY:
The purpose of this study is to determine safety and efficacy of 30mg daily dose of clevudine (L-FMAU) at 24 weeks of treatment in chronic HBV infected patients with HBeAg negative

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were between 18 and 60, inclusive
2. Patients with HBV DNA levels 1 x 105 copies/mL within 30 days of baseline.
3. Patients who were documented to be HBsAg positive for > 6 months (documentation of positive HBsAg for the previous 6 months included previous laboratory reports showing HBsAg positive at least 6 month ago OR lab results showing IgM anti-HBc negative and IgG anti-HBc positive at screening).
4. Patients who were HBeAg negative and HBeAb positive.
5. Patients with ALT levels which were in the range of ≥1.2 and < 15 times the upper limit of normal (ULN) and bilirubin levels less than 2.0 mg/dL, prothrombin time of less than 1.7 (INR), a serum albumin level of at least 3.5 g/dL.
6. Women of childbearing potential with a negative serum (β-HCG) pregnancy test taken within 14 days of starting therapy.
7. Patients who were able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patients who were currently receiving antiviral, immunomodulatory or corticosteroid therapy.
2. Patients previously treated with lamivudine, lobucavir, famciclovir, adefovir or any other investigational nucleoside for HBV infection. Previous treatment with interferon that had ended less than 6 months prior to the screening visit.
3. Patients with a history of ascites, variceal hemorrhage or hepatic encephalopathy.
4. Patients coinfected with HCV, HDV or HIV.
5. Patients with clinical evidence of liver mass or with alfa-fetoprotein > 50 ng/mL
6. Patients who were pregnant or breast-feeding.
7. Patients who were unwilling to use an "effective" method of contraception during the treatment period and for up to 3 months after cessation of therapy. For males, condoms should be used. Females had to be surgically sterile (via hysterectomy or bilateral tubal ligation) or post-menopausal or using at least medically acceptable barrier method of contraception (i.e. IUD, barrier methods with spermicide or abstinence)
8. Patients with a clinically relevant history of abuse of alcohol or drugs.
9. Patients with a significant gastrointestinal, renal, hepatic (decompensated), broncho-pulmonary, biliary diseases except asymptomatic GB stone, neurological, cardiovascular, oncologic or allergic disease. The patient with a benign tumor was excluded if judged by an investigator that the continuation of study would be interfered by benign tumor.
10. Patients with creatinine clearance less than 60mL/min as estimated by the following formula:

(140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80
Dates: Start 2003-07; Study Completion 2004-12

PRIMARY OUTCOMES:
Efficacy:
Antiviral activity (change from baseline in HBV DNA (log 10))
Safety:
Laboratory tests
Adverse Events
Vital signs
ECG

SECONDARY OUTCOMES:
Efficacy
Antiviral activity: proportion of patients with HBV DNA below the assay limit of detection (<4,700 copies/mL by Digene Hybrid Capture II assay)
Biochemical improvement (e.g. ALT normalization )

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Suk Lee, MD. PhD, Principal Investigator — Seoul National University Hospital
Locations (30):
- South Korea (30):
  - St. Mercy's Hospital, Bupyoung-dong, Bupyoung-gu, Incheon
  - Pusan Paik Hospital, Gaegeum-dong, Busan
  - Kangbuk Samsung Hospital, Pyoung-dong, Chongro-gu, Seoul
  - Keimyumg University Dongsan Medical Center, Jung-gu, Daegu
  - Chonnam National University Hospital, Hak-1-dong, Dong-gu, Gwangju-si
  - Korea University Guro Hospital, Seoul, Guro-gu
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Seoul National University Hospital, Seoul, Jongno-Gu
  - Inha University Hospital, Sinhŭng-dong, Jung-gu, Incheon
  - Seoul Asan Medical Center, Pungnap-dong, Kangnam-gu, Seoul
  - Yongdong Severance Hospital, Togok-tong, Kangnam-gu, Seoul
  - St. Holly Family Mary's Hospital, Bucheonae, Kyounggi-do
  - National Cancer Center, Ilsan-gu, Kyounggi-do
  - Pochon CHA University Hospital, Seongnam-gu, Kyounggi-do
  - Yeungnam University Medical Center, Dae Myoung-dong, Nam-gu, Taegu
  - Gil Medical Center, Incheon, Namdong-Gu
  - Nowon Eulji Hospital, Hagyeil-tong, Nowon-gu, Seoul
  - St. Vincent's Hospital, Chi-dong, Paldal-gu, Suwon
  - Pusan National University Hospital, Ami-dong, Seo-gu, Pusan
  - Kosin Medical Center, Amnam-dong, Seo-gu, Pusan
  - KangNam St. Mary's Hospital, Banpo-dong, Seocho-gu, Seoul
  - Severance Hospital, Shinchon- Dong, Seodaemun-gu, Seoul
  - Seoul Paik Hospital, Jeo-dong, Seoul
  - Samsung Medical Center, Ilwon-dong, Songpa-gu, Seoul
  - Korea University Anam Hospital, Anam-dong, Sungbuk-ku, Seoul
  - Ehwa Womans University Mokdong Hospital, Mokdong, Yangcheon-gu, Seoul
  - Kangnam Sacred Heart Hospital, Daelim-dong, Yongdeungpo-gu, Seoul
  - Soon Chun Hyang University Hospital, Hannam-dong, Yongsan-gu, Seoul
  - St. Mary's Hospital, Seoul, Yungdungpo-Gu

REFERENCES:
- [Derived] Yoo BC, Kim JH, Kim TH, Koh KC, Um SH, Kim YS, Lee KS, Han BH, Chon CY, Han JY, Ryu SH, Kim HC, Byun KS, Hwang SG, Kim BI, Cho M, Yoo K, Lee HJ, Hwang JS, Kim YS, Lee YS, Choi SK, Lee YJ, Yang JM, Park JW, Lee MS, Kim DG, Chung YH, Cho SH, Choi JY, Kweon YO, Lee HY, Jeong SH, Yoo HW, Lee HS. Clevudine is highly efficacious in hepatitis B e antigen-negative chronic hepatitis B with durable off-therapy viral suppression. Hepatology. 2007 Oct;46(4):1041-8. doi: 10.1002/hep.21800. PMID 17647293